CLINICAL TRIAL: NCT02897336
Title: Ultrasound-guided Caudal or Interlaminar Injection? A Comparative Study of Epidural Corticosteroid Injections in the Treatment of Lumbar Disk Herniation-related Sciatica
Brief Title: Ultrasound-guided Caudal or Interlaminar Corticosteroid Epidural Injection for Sciatica
Acronym: HiatUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A01502-47
Record Dates: First submitted 2016-08-31; First posted 2016-09-13 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Sciatica
MeSH Terms: conditions — Sciatica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultrasound-guided (Experimental): ultrasound-guided caudal epidural corticosteroid injection
  Interventions: Procedure: ultrasound-guided
- interlaminar (Active Comparator): interlaminar epidural corticosteroid injection
  Interventions: Procedure: interlaminar

INTERVENTIONS:
Procedure: ultrasound-guided — ultrasound-guided caudal epidural corticosteroid injection
  Arms: ultrasound-guided
Procedure: interlaminar — interlaminar epidural corticosteroid injection
  Arms: interlaminar

SUMMARY:
An open-label randomized trial to compare the efficacy of ultrasound-guided caudal and interlaminar corticosteroid injections for the treatment of lumbar disk herniation-related sciatica.

DETAILED DESCRIPTION:
An open-label randomized trial conducted in one centre to compare the efficacy of ultrasound-guided caudal and interlaminar corticosteroid injections for the treatment of lumbar disk herniation-related sciatica. 30 male and female patients will be included in each group. The primary outcome measure will be a 30% decrease in lower limbs pain as assessed by a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* radicular pain (sciatica or cruralgia) for more than 2 weeks
* failure of analgesics and NSAIDs
* without neurological deficiency (motor weakness lower or equal to 3/5)
* a lumbar disk herniation on MRI or CT dating less than 3 months

Exclusion Criteria:

* history of lumbar surgery
* history of epidural injection during the last 3 months
* radicular pain not due to disk herniation
* a contraindication to epidural injection (infection, diabetes)
* history of allergic reaction to corticosteroid
* patient under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
lower limbs pain | day 15
  a 30% decrease in lower limbs pain using a visual analog scale

SECONDARY OUTCOMES:
Oswestry questionnaire | day 15 - month 1 - month 3 - month 6
  low back pain disability assessment using Oswestry questionnaire
A decrease of radicular pain with a pain numerical scale lower or equal to 3/10 | day 15 - month 1 - month 3 - month 6
  pain numerical scale lower or equal to 3/10
neurological deficiency assessed by neurological examination | day 15 - month 1 - month 3 - month 6
  motor weakness or sensitive deficiency in lower limbs
drugs | day 15 - month 1 - month 3 - month 6
  decrease in analgesic treatment
medical outcome | day 15 - month 1 - month 3 - month 6
  Medical Outcome study Short Form (SF-36)
resumption of work | day 15 - month 1 - month 3 - month 6
  deadline of resumption of work
number of patients with treatment-related adverse events as assessed by CTCAE v4.0 | day 15 - month 1 - month 3 - month 6
  adverse events assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No